CLINICAL TRIAL: NCT05213728
Title: A Phase 1, Open-label, Safety and Immunogenicity Study of an Oral Multi-dose Administration Regimen With an Adenoviral-vector Based Tablet Norovirus Vaccine (VXA-G1.1-NN) Expressing GI.1 VP1 Administered to Healthy Adult Volunteers
Brief Title: A Phase 1, Open-label, Safety and Immunogenicity Study of an Oral Multi-dose Administration Regimen With an Adenoviral-vector Based Tablet Norovirus Vaccine (VXA-G1.1-NN) Administered to Healthy Adult Volunteers
Acronym: (VXA-G1-1-NN)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VXA-NVV-106
Record Dates: First submitted 2022-01-18; First posted 2022-01-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2022-09

CONDITIONS: Norovirus Infections
MeSH Terms: conditions — Caliciviridae Infections

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort 1 (Experimental): Single 1E11 dose administered via multiple sub-doses over a 4-hour period in adults (18-55 yrs).
  Interventions: Biological: VXA-G1.1-NN

INTERVENTIONS:
Biological: VXA-G1.1-NN — Norovirus GI.1 Norwalk VP1 Vaccine (VXA-G1.1-NN) E1/E3-Deleted Replication-Defective Recombinant Adenovirus 5 with Adjuvant Oral Tablet Vaccine.
  Other Names: Oral Tableted Ad5 Norovirus GI.1 Vaccine

SUMMARY:
Subjects will receive multiple sub-doses over a 4-hour period to deliver a total overall dose of 1E11. Evaluations of immunogenicity, safety, and tolerability will be evaluated. The active period consists of data collection at Day 1, Day 8, and Day 29. Safety follow-up continues by phone screen at Day 180 and Day 365.

DETAILED DESCRIPTION:
Primary Objective

* To determine the immunogenicity of the VXA-G1.1-NN oral vaccine administered via multiple sub-doses over a 4-hour period to deliver a total dose of

  1E11 IU ±0.5 log Secondary Objectives
* To determine the safety and tolerability of the VXA-G1.1-NN oral vaccine administered via multiple sub-doses over a 4-hour period to deliver a total dose of 1E11 IU ±0.5 log

This is an open-label study in healthy adult participants aged 18-55 years old. The study will enroll 8 subjects to a single treatment cohort, all of whom will receive a single 1E11 IU± 0.5 log at Day 1. This dose will be administered in a step wise manner over 4 hours with 1/3 of the dose administered at T=0, 1/3 of the dose administered at T= 2 hours and 1/3 of the dose administered at T=4 hours.

The study will include a Screening Period, Active Period (Day 1 to Day 29, 4 weeks post vaccination) and a Safety Follow-up Period through 12 months post vaccination (Day 365). In addition, participants will be contacted by phone during the Safety Follow-up Period to assess for Serious Adverse Events (SAEs), AEs of Special Interest (AESIs) and New Onset of Chronic Illness (NOCIs).

After signing an informed consent, participants will undergo screening assessments to determine study eligibility within a 30-day screening period. Eligible participants will be enrolled and receive their first dose of study vaccine on Day 1.

During the Active Period, participants will record any potential solicited symptoms of reactogenicity daily for 1 week post study vaccination. Participants will return to the site as specified in the Schedule of Activities to have safety assessments and samples collected for evaluation of immunogenicity. Approximately 8 subjects will be vaccinated in the active phase.

The following study visits and remote contacts will be conducted during the study:

Active Period:

* Screening Period (Days -30 to -1)
* Day 1 Visit (Baseline assessments, vaccination, sample collection)
* Day 8 Visit (Safety assessments, sample collection)
* Day 29 End of Active Period; (Safety assessments, sample collection)

Safety Follow-Up Period:

* Day 180 (follow-up phone call for safety)
* Day 365 (follow-up phone call for safety): Study completion

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years old, inclusive, at day of signing Informed Consent Form (ICF)
2. General good health, without significant uncontrolled medical illness, based on medical history, physical examination, vital signs, and clinical laboratories (CBC, chemistry, and urinalysis) as determined by the investigator in consultation with the Research Monitor and Sponsor
3. Body mass index (BMI) between 17 and 35 kg/m2 at screening
4. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol
5. Available for all planned visits and phone calls, and willing to complete all protocol-defined procedures and assessments (including ability and willingness to swallow multiple small enteric-coated tablets per study dose)
6. Female participants must provide a negative pregnancy test at each required visit and fulfill one of the following criteria:

   1. At least 1 year post-menopausal (defined as amenorrhea for ≥12 consecutive months prior to Screening without alternative medical cause)
   2. Surgically sterile
   3. Use of oral, implantable, transdermal or injectable contraceptives for 30 days prior to initial vaccination and until 60 days after the last vaccination. The form of contraception must be approved by the Investigator
   4. A reliable form of contraception must be approved by the Investigator (e.g., double barrier method, Depo-Provera, intrauterine device, Norplant, oral contraceptives, contraceptive patches)
   5. Not be sexually active (abstinent) or be in a relationship with partner who is sterile (must be discussed with site staff and documented)
7. Male participants must agree not to father a child or donate sperm, as well as to use contraception/barrier (a male condom) or be abstinent from heterosexual intercourse during the study active period (Day 29)

Exclusion Criteria:

1. Presence of significant uncontrolled medical or psychiatric illness (acute or chronic) including institution of new medical/surgical treatment or significant dose alteration for uncontrolled symptoms or drug toxicity within 3 months of screening and reconfirmed at baseline
2. Cancer, or received treatment for cancer, within past 3 years (excluding basal cell carcinoma or squamous cell carcinoma)
3. Presence of immunosuppression or medical condition possibly associated with impaired immune responsiveness, including diabetes mellitus 1 and 2
4. History of irritable bowel disease or other inflammatory digestive or gastrointestinal condition that could affect the distribution/safety evaluation of an orally administered vaccine targeting the mucosa of the small intestine Norwalk GI.1 (VXA-G1.1-NN) Protocol No. VXA-NVV-106

   ________________________________________________________________________________

   _________________________________________________________________________________ Version 1.2 Confidential Page 11 of 42 Date: 04 Jan 2022

   Such conditions may include but are not limited to:
   1. Esophageal Motility Disorder
   2. Malignancy
   3. Malabsorption
   4. Pancreaticobiliary disorders
   5. Irritable bowel syndrome
   6. Inflammatory Bowel Disease
   7. Surgical Resection
   8. GERD
   9. Hiatal Hernia
   10. Peptic Ulcer (History of cholecystectomy is not exclusionary)
5. History of any form of angioedema
6. History of serious reactions to any vaccination such as anaphylaxis, respiratory problems, hives or abdominal pain
7. Diagnosed bleeding disorder or significant bruising or bleeding difficulties that could make blood draws problematic
8. Any condition that resulted in the absence or removal of the spleen
9. Acute disease within 72 hours prior to vaccination defined as the presence of a moderate or severe illness (as determined by the Investigator through medical history and physical exam); assessment may be repeated during screening period
10. Presence of a fever ≥ 38oC measured orally at baseline; assessment may be repeated during screening period
11. Laboratory values outside the range of normal for platelet counts and the following coagulation tests: PT/INR, aPTT and fibrinogen
12. Any of the following history or conditions that may lead to higher risk of clotting events and/or thrombocytopenia:

    1. Family or personal history of bleeding or thrombosis
    2. History of heparin-related thrombotic events, and/or receiving heparin treatments
    3. History of autoimmune or inflammatory disease
    4. Presence of any of the following conditions known to increase risk of thrombosis within 6 months prior to screening:

       * Recent surgery other than removal/biopsy of cutaneous lesions
       * Immobility (confined to bed or wheelchair for 3 or more successive days)
       * Head trauma with loss of consciousness or documented brain injury
       * Receipt of anticoagulants for prophylaxis of thrombosis
       * Recent clinically significant infection
13. Any significant hospitalization within the last year which in the opinion of Norwalk GI.1 (VXA-G1.1-NN) Protocol No. VXA-NVV-106
14. Any other condition that in the clinical judgment of the investigator would jeopardize the safety or rights of a participant taking in the study, would render the participant unable to comply with the protocol or would interfere with the evaluation of the study endpoints
15. Positive human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV) tests at screening visit
16. Positive urine drug screen for drugs of abuse at screening
17. Positive breath or urine alcohol test at screening and baseline
18. Receipt of a licensed vaccine within 14 days prior to baseline vaccination or planned administration during the study active period
19. Use of antibiotics, proton pump inhibitors, H2 blockers or antacids within 7 days prior to study drug administration or planned use during the active study period
20. Use of medications known to affect the immune function (e.g., systemic corticosteroids and others) within 2 weeks before study vaccination or planned use during the active period
21. Daily use of nonsteroidal anti-inflammatory drugs within 7 days prior to study vaccination or planned use during the active study period
22. Administration of any investigational vaccine, drug or device within 8 weeks preceding study vaccination (Day 1), or planned use within the duration of the study
23. Donation or use of blood or blood products within 30 days prior to study vaccination or planned donation during the active study period
24. History of drug, alcohol or chemical abuse within 1 year of screening
25. History of hypersensitivity or allergic reaction to any component of the investigational vaccine, including but not limited to fish gelatin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Rate of Solicited Symptoms of Reactogenicity | Up to Day 8
  To assess the safety and tolerability of an oral tableted vaccine by collection of solicited symptoms of vaccine reactogenicity recorded daily using a subject diary card for 1 week post initial vaccination at Day 1.
To assess the induction of VP1-specific Immunoglobin A (IgA) antibody-secreting cells (ASC) by ELISpot assay | Change from baseline at Day 8
  Change from baseline in VP1-specific Immunogolobin A (IgA) antibody-secreting cells (ASC) by ELISpot assay will be evaluated at Day 8
To assess histo-blood group antigen (HBGA) blocking antibodies by blockade titer (BT50) | Change from baseline at Day 29
  Change from baseline in histo-blood group antigen (HBGA) blocking antibodies evaluated at Day 29
To assess VP1-specific serum Immunoglobin G (IgG) by Mesoscale Discovery (MSD) assay | Change from baseline at Day 29
  Change from baseline in VP1-specific Immunoglobin G (IgG) by Mesoscale Discovery (MSD) assay will be evaluated at Day 29
To assess the VP1-specific serum Immunoglobin A (IgA) by Mesoscale Discovery (MSD) assay | Change from baseline at Day 29
  Change from baseline in VP1-specific serum IgG by Mesoscale Discovery (MSD) will be evaluated at Day 29

CONTACTS AND LOCATIONS:
Overall Officials: James Cummings, MD, Study Director — Vaxart, Inc.
Locations (1):
- AltaSciences LA, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No